CLINICAL TRIAL: NCT05071508
Title: Ability of Bedside Ultrasound to Predict and Optimize Metabolic and Neurodevelopmental Outcomes in Premature Infants in the Neonatal Intensive Care Unit
Brief Title: US and Neurodevelopmental Outcomes in the Neonatal Intensive Care Unit (NICU)
Status: Completed | Type: Observational
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Other Study IDs: PEDS-2020-28483
Record Dates: First submitted 2019-12-20; First posted 2021-10-08 (Actual); Last update posted 2025-02-06 (Actual); Status verified 2025-02

CONDITIONS: Premature Birth
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Preterm Infants: Premature infants (born between 25 and 34 + 6 weeks gestational age) admitted to the University of Minnesota Masonic Children's Hospital NICU

SUMMARY:
The objective of the project is to identify clinical factors (nutritional and non-nutritional) which are associated with ultrasound measurements of muscle and adipose tissue and to determine whether these ultrasound measurements are predictive of later metabolic and neurodevelopmental outcomes in premature infants, a population at risk for developmental delay, obesity, and metabolic disease. The investigators expect that a better understanding of these relationships will lead to the incorporation of ultrasound into routine nutritional management of preterm infants and allow for future optimization of their overall health and development.

DETAILED DESCRIPTION:
The specific aims are as follows:

1. To identify clinical factors that are associated with muscle and adipose tissue measurements. The investigators will examine the relationship between clinical factors such as calorie and protein intake during hospitalization, days on parenteral nutrition, C-Reactive Protein and other clinical surrogates for inflammation and both muscle and adipose tissue measured bi-weekly using bedside ultrasound. The investigators will collect anthropometric and ultrasound measurements bi-weekly and whole body composition (utilizing ADP) data at 35 weeks postmenstrual age (PMA)/discharge from the Neonatal Intensive Care Unit. All other clinical data will be collected throughout the hospital stay.
2. To determine whether muscle thickness and cross-sectional area are predictive of improved neurodevelopmental outcomes. The investigators will assess the relationship between ultrasound measurements of muscle with neurodevelopmental outcomes at 35 weeks PMA/discharge and 4 months corrected age. The investigators will utilize Event Related Potentials (ERP) to measure speed of processing and recognition memory as early markers of brain development.
3. To determine whether measurements of adipose tissue are predictive of later adverse metabolic outcomes. The investigators will assess the relationship between adipose tissue thickness and blood pressure and total body adiposity (using air-displacement plethysmography) at 35 weeks PMA/discharge and 4 months corrected age.

ELIGIBILITY:
Inclusion Criteria:

* preterm infants born between 25 and 34+6 weeks gestation admitted to University of Minnesota Masonic Children's Hospital Neonatal Intensive Care Unit
* medically stable at time of air displacement measurements

Exclusion Criteria:

* infants that require medical support preventing ADP measurements from being taken

Ages: 25 Weeks to 34 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Preterm infants
Sampling Method: Non-Probability Sample
Enrollment: 37 (Actual)
Dates: Start 2020-02-20 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Blood pressure at 35 weeks | 35 weeks corrected age
  blood pressure (systolic and diastolic)
Blood pressure at 4 mo | 4 months corrected age
  blood pressure (systolic and diastolic)
Weight data inpatient | 35 weeks corrected age
  weight in kg
Length data inpatient | 35 weeks corrected age
  length in cm
Weight data outpatient | 4 months corrected age
  weight in kg
Length data outpatient | 4 months corrected age
  length in cm
Fat mass inpatient | 35 weeks corrected age
  fat mass (kg)
Fat-free mass inpatient | 35 weeks corrected age
  fat-free mass (kg)
Percent body fat inpatient | 4 months corrected age
  percent body fat (kg/kg)
Fat mass outpatient | 4 months corrected age
  fat mass (kg)
Fat-free mass outpatient | 4 months corrected age
  fat-free mass (kg)
Percent body fat outpatient | 4 months corrected age
  percent body fat (kg/kg)
Ultrasound adipose measures inpatient | 35 weeks corrected age
  adipose tissue (cm)
Ultrasound muscle measures inpatient | 35 weeks corrected age
  muscle thickness (cm)
Ultrasound adipose measures outpatient | 4 months corrected age
  adipose tissue (cm)
Ultrasound muscle measures outpatient | 4 months corrected age
  muscle measurements (cm)
ERP data inpatient | 35 weeks corrected age
  ERP paradigm
ERP data outpatient | 4 months corrected age
  ERP paradigms

CONTACTS AND LOCATIONS:
Overall Officials: Sara E Ramel, MD, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No